CLINICAL TRIAL: NCT05959252
Title: BivaLirudin versUS Heparin in ECMO - A Registry-embedded, Randomised, Open Label, Feasibility Trial Comparing Two Anticoagulation Strategies in Patients on Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: BivaLirudin versUS Heparin in Extracorporeal Membrane Oxygenation
Acronym: BLUSH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sydney Local Health District (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/ETH00443
Record Dates: First submitted 2023-07-02; First posted 2023-07-25 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Extracorporeal Membrane Oxygenation Complication
Keywords: ECMO; Bivalirudin; Heparin; Extracorporeal membrane oxygenation
MeSH Terms: interventions — Heparin; bivalirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bivalirudin (Active Comparator): Bivalirudin protocol with target activated thromboplastin time (aPTT) of 50-70 seconds
  Interventions: Drug: Bivalirudin
- Unfractionated Heparin (Active Comparator): Unfractionated heparin protocol with target anti-Xa of 0.3-0.5 IU/mL
  Interventions: Drug: Unfractionated heparin

INTERVENTIONS:
Drug: Unfractionated heparin — Unfractionated Heparin protocol with target anti-Xa of 0.3-0.5 IU/mL
  Other Names: Heparin
  Arms: Unfractionated Heparin
Drug: Bivalirudin — Bivalirudin protocol with target aPTT 50-70 seconds
  Arms: Bivalirudin

SUMMARY:
The goal of this open label randomised clinical trial is to compare Bivalirudin versus Heparin for anticoagulation in patients requiring extracorporeal membrane oxygenation support.

The main question it aims to answer are include the ability to maintain anticoagulation within defined therapeutic range, bleeding and thrombotic complications and a comparison of the total cost of anticoagulation care.

Participants will be randomised to either anticoagulation with Bivalirudin or anticoagulation with Unfractionated Heparin.

DETAILED DESCRIPTION:
Rationale:

Anticoagulation whilst on extracorporeal membrane oxygenation (ECMO) is required. Bleeding and thrombotic complications whilst on ECMO are common and may effect the patient outcome. The optimal anticoagulant for ECMO patients is not clear and there exists no randomised control trial data comparing anticoagulants on ECMO. This Phase 2b trial will provide data to enable larger definitive phase III trials to determine the best anticoagulant whilst on ECMO.

Hypothesis: Hypothesis: In adults ECMO patients'; anticoagulation with Bivalirudin results in more samples within therapeutic range than unfractionated Heparin. Total anticoagulation costs with Bivalirudin are similar to unfractionated Heparin.

The objectives of this study is to assess anticoagulation protocol of bivalirudin versus unfractionated heparin and assess the to the cost of each protocol.

ELIGIBILITY:
INCLUSION CRITERIA

* Patients receiving ECMO
* Age: 18 years or older
* Ability to randomise the patient within 4 hours of ECMO support initiation

EXCLUSION CRITERIA

* Post-cardiotomy ECMO patients
* Contraindication to heparin or bivalirudin at time of randomisation e.g., active bleeding
* Heparin induced thrombotic thrombocytopenia syndrome
* Where the patient is expected to be disconnected from ECMO in the next day after cannulation.
* Limitations of care put in place either through patient wishes or the treating medical teams
* Other reason where the treating physician deems the study is not in the patient's best interest
* Patients who are suspected or confirmed to be pregnant
* Inherited bleeding or thrombotic disorders, Systemic Lupus Erythematosus patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Time in therapeutic range | 30 days
  Proportion of monitoring samples within therapeutic range

SECONDARY OUTCOMES:
Enrolment rate | 30 days
  Enrolment rate
Reasons for non-enrolment | 30 days
  Reasons for non-enrolment of eligible patients into the study
Crossover between arms | 30 days
  The number of cross over patients between arms of the study
Circuit changes | 30 days
  The number of circuit changes and length of circuit life
Daily mean aPTT and anti-Xa | 30 days
  Daily mean aPTT and anti-Xa versus stated range
Serious adverse events (SAEs) | 30 days
  Number of SAEs
Protocol violations | 30 days
  Number of protocol violations
Thrombotic events | 30 days
  Number of deep vein thrombosis identified by ultrasound or CT
Major bleeding events defined by International Society of Thrombosis and Haemostasis (ISTH) | 30 days
  Major bleeding was defined according to the criteria as clinically overt bleeding which was fatal or associated with any of the following: (a) a fall in hemoglobin level of 2 g/dL or more or documented transfusion of at least 2 units of packed red blood cells, (b) involvement of a critical anatomical site (intracranial, spinal, ocular, pericardial, articular, intramuscular with compartment syndrome, retroperitoneal)
Bleeding events defined by Bleeding Academic Research Consortium (BARC) | 30 days
  Number of bleeding events as per BARC
  Hemorrhagic complications assessed and adapted as per Bleeding Academic Research Consortium (BARC) Type 0: No bleeding Type 1: Bleeding requiring transfusion of packed red blood cells (PRBC) or reduction of unfractionated heparin Type 2: Bleeding requiring transfusion of PRBC and reduction of unfractionated heparin Type 3: Life-threatening bleeding requiring, transfusion of PRBC, surgical intervention or discontinuation of ECMO Type 4: Any fatal bleeding
Survival to Intensive care Unit (ICU) discharge | 30 days
  Survival to discharge from ICU (percentage of patients surviving to ICU discharge)
Survival to hospital discharge | 30 days
  Hospital Survival (percentage of patients surviving hospital discharge)
Blood product usage | 30 days
  Total amount of red blood cells (RBC), platelets, plasma and blood products used during extracorporeal membrane oxygenation support
Cost | 30 days
  Total cost of of extracorporeal membrane oxygenation support that includes blood products, blood tests and complications (measured in United States dollars)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Prince Alfred Hospital, Sydney, New South Wales, Australia